| <b>Participant</b> | ID: | | |
|--------------------|-----|---|-------|
| | | - | <br>- |





Implementation studio, an innovative, structured approach to facilitate rural community-based organizations' adaptation and implementation of evidence-based interventions

## Community-based Organization (CBO) Client Verbal Consent Script

Dr. Linda Ko, PhD Principal Investigator, Associate Member Fred Hutchinson Cancer Research Center

Email: <u>lko@fredhutch.org</u> Phone: (206) 667-7182 Geno Ibarra
Project Manager
Center for Community Health Promotion

Email: <a href="mailto:gibarra@fredhutch.org">gibarra@fredhutch.org</a> Phone: (509) 837-6359

Follow this script to consent the CBO's clients/participants to participant in the research project. This procedure is applicable for both incoming and outgoing calls. When contacting a participant, follow the steps and document the information as indicated on the participant contact log. Prior to the call, review the participant contact log for the participant's name and pertinent information.

#### **OUTGOING CALLS:**

**IF YOU REACH VOICEMAIL:** This is [STAFF MEMBER NAME] calling on behalf of [CBO's NAME] and the [PROJECT NAME]. I am trying to reach [PARTICPANT NAME] to confirm participation in a research project. Please call me back at [PHONE NUMBER] to schedule a time to talk. Thank you.

**IF THE CALL IS ANSWERED:** Hello, I'm [STAFF MEMBER NAME] calling on behalf of [CBO's NAME] and the [PROJECT NAME]. Is [PARTICPANT NAME] available to talk?

IF NO: Okay. Please have [PARTICIPANT NAME] call me back at [PHONE NUMBER]. Thank you.

IF YES (SPEAKING TO PARTICIPANT): Good day is this [PARTICPIANT NAME]? CONFIRM YOU ARE SPEAKING WITH PARTICIPANT BY VERIFYING NAME

**IF YES – CONTINUE WITH SCRIPT:** I'm reaching out today to because you expressed interest in participating in research project on behalf of [PROJECT NAME] and a team of researchers at the Fred Hutchinson Cancer Research Center, a program called Implementation Studio. The purpose of this program is to help community-based organizations implement interventions that are known to be successful in helping people get screened for cancer. A community-based organization in your community is participating in the Implementation Studio. We want to see if the interventions help clients of this community-based organization, like you, get screened for cancer. This study will help us understand how to improve the program so that it is relevant to your community.

If you decide to take part in this study, we will ask you to participate in a phone interview about the cancer screening program to be implemented in your community.

- First, we will ask you to participate in a phone survey where we will ask you some questions about your demographics to determine if you are eligible to participate in the study. This call will take about 15 minutes.
- Then, you will participate in a phone interview where we will ask about how to optimize the cancer screening intervention for cultural relevance and acceptability in your community. The interview will take about 30 minutes. You will receive \$10 for participating in the interview.
- You will then have the opportunity to participate in the cancer screening program provided by the community-based organization. We will ask you to complete a survey before and after you receive the program. The survey will ask you about your demographics, access to healthcare, knowledge and

| <b>Participant</b> | :ID: |
|--------------------|------|
| Participani | : טו |

beliefs about cancer screening, and your experience in the program. You will receive \$20 for participating in the program and surveys.

There are no costs to you for participating in this study. You will receive up to \$30 for participating in the study.

Participation of the organization's clients will help us develop the Implementation Studio into a useful tool for the community-based organization. Client feedback will help the research team and the organization how to adapt the cancer screening interventions for rural communities. Ultimately, this will help increase access to evidence-based health programs in rural communities.

We do not anticipate any risks or trouble to you for participating in the study. However, answering questions about your personal viewpoint regarding the intervention may make you feel uncomfortable.

Your participation in this study is voluntary. You may choose not to answer any questions that make you feel uncomfortable and you may refuse to participate at any time. There is no right or wrong answer in the interviews; we just want to know your opinions and have your participation. There is no penalty or loss of benefits to you if you choose to stop your participation.

Everything you say in this study is private and will not be shared with anyone outside the research team. Reported or published data will not identify anyone by name or other personal information. To protect your privacy, project staff will give each participant an identification (ID) number. Information linking the participant name and study ID number is kept in a password protected computer file. Project staff will destroy all study materials with personal information three years after the study has been completed. This includes permanently deleting the audio recording of the interviews at the conclusion of the study and shredding the signed consent forms. All shredded paper will be placed in a private recycling bin. By law, the Institutional Review Board (IRB) at FHCRC may ask to look at participant data. An IRB is a group that reviews the study to protect your rights as a research participant.

If you have questions or complaints about the research study you may I can clarify questions for you know, or I can provide you with the phone numbers of the Principal Investigator, Linda Ko or Community Project Manager, Genoveva Ibarra. Both speak Spanish and English. If you have any questions about the interview today and the overall research, or your rights as a research participant, you may contact the Fred Hutch Institutional Review office. I can provide you with that number.

Do you have any questions regarding the focus group or the research project?

#### IF YES - ANSWER QUESTIONS AND PROVIDE APPROPRIATE PHONE NUMBERS:

PI: Dr. Linda Ko (206) 667-7182 Project Manager: Genoveva Ibarra (509) 837-6359

IRB: Director of Institutional Review Office (206) 667-5900

### IF NO - PROCEED TO NEXT STATEMENT

Are you in agreement with the consent that I read?

# IF YES – PROCEED TO NEXT STATEMENT IF NO – THANK PARTICIPANT FOR THEIR TIME AND END CALL

Since you agree with the consent that I have read, can we proceed with participation in the study as outlined?

IF YES – PROCEED TO INTERVIEW QUESTIONS
IF NO – THANK PARTICIPANT FOR THEIR TIME AND END CALL

FHCRC IRB Approval

07/22/2020

Document Release Date

CBO Client Verbal Consent Vrs. 1 IR File 10307 IRB Approved: XX/XX/2020 Page 2 of 2